CLINICAL TRIAL: NCT01835431
Title: A Trial Investigating the Efficacy and Safety of Insulin Degludec/Insulin Aspart Once Daily Plus Insulin Aspart for the Remaining Meals Versus Insulin Detemir Once or Twice Daily Plus Meal Time Insulin Aspart in Children and Adolescents With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN5401-3816; 2012-003566-41 (EudraCT Number); U1111-1133-0958 (Other: WHO); PIP no. be confirmed (Other: EMA)
Record Dates: First submitted 2013-04-16; First posted 2013-04-19 (Estimated); Results first posted 2015-11-17 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec, insulin aspart drug combination; Insulin Aspart; Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin degludec/insulin aspart (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart; Drug: insulin aspart
- Insulin detemir (Active Comparator)
  Interventions: Drug: insulin detemir; Drug: insulin aspart

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — Administered subcutaneously (s.c., under the skin) once daily with a main meal. Dose individually adjusted.
  Arms: Insulin degludec/insulin aspart
Drug: insulin aspart — Administered s.c. with the remaining meals. Dose individually adjusted.
  Arms: Insulin degludec/insulin aspart
Drug: insulin detemir — Administered s.c. once or twice daily. Dose individually adjusted. Subjects will continue with their pre-trial dosing scheme (once (OD) or twice daily (BID)) and will be allowed to switch from OD to BID dosing.
  Arms: Insulin detemir
Drug: insulin aspart — Administered s.c. at meal-times. Dose individually adjusted.
  Arms: Insulin detemir

SUMMARY:
This trial is conducted in Asia, Europe and North and South America. The aim of the trial is to investigate the efficacy and safety of insulin degludec/insulin aspart once daily plus insulin aspart for the remaining meals in children and adolescents with type 1 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria: - Informed consent obtained before any trial related activities. Trial related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial - Subjects diagnosed with type 1 diabetes mellitus - HbA1c below or equal to 11.0% Exclusion Criteria: - Known hypoglycaemic unawareness or recurrent severe hypoglycaemic events as judged by the investigator - More than 1 episode of diabetic ketoacidosis requiring hospitalisation within the last 3 months prior to Visit 1 (Screening) - Any chronic disorder or significant concomitant disease, which in the investigator's opinion might jeopardise the subject's safety or compliance with the protocol

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 362 (Actual)
Dates: Start 2013-10-17 (Actual); Primary Completion 2014-11-07 (Actual); Study Completion 2014-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (65):
- United States (22):
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Sacramento, California
  - Novo Nordisk Investigational Site, Aurora, Colorado
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Maitland, Florida
  - Novo Nordisk Investigational Site, Melbourne, Florida
  - Novo Nordisk Investigational Site, Tallahassee, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Idaho Falls, Idaho
  - Novo Nordisk Investigational Site, Springfield, Illinois
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Worcester, Massachusetts
  - Novo Nordisk Investigational Site, Kansas City, Missouri
  - Novo Nordisk Investigational Site, Buffalo, New York
  - Novo Nordisk Investigational Site, Tulsa, Oklahoma
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Dallas, Texas
- Belgium (2):
  - Novo Nordisk Investigational Site, Brussels
  - Novo Nordisk Investigational Site, Leuven
- Brazil (3):
  - Novo Nordisk Investigational Site, Curitiba, Paraná
  - Novo Nordisk Investigational Site, Porto Alegre, Rio Grande do Sul
  - Novo Nordisk Investigational Site, São Paulo, São Paulo
- Canada (4):
  - Novo Nordisk Investigational Site, Vancouver, British Columbia
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Mississauga, Ontario
  - Novo Nordisk Investigational Site, Montreal, Quebec
- Novo Nordisk Investigational Site, Zagreb, Croatia
- Czechia (3):
  - Novo Nordisk Investigational Site, Olomouc
  - Novo Nordisk Investigational Site, Pardubice
  - Novo Nordisk Investigational Site, Prague
- India (5):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, New Dehli, New Delhi
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
- Israel (6):
  - Novo Nordisk Investigational Site, Beersheba
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Tel Aviv
  - Novo Nordisk Investigational Site, Tel Litwinsky
  - Novo Nordisk Investigational Site, Ẕerifin
- Novo Nordisk Investigational Site, Skopje, North Macedonia
- Poland (2):
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Warsaw
- Russia (5):
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Tomsk
  - Novo Nordisk Investigational Site, Ufa
- Serbia (3):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Niš
  - Novo Nordisk Investigational Site, Novi Sad
- Novo Nordisk Investigational Site, Ljubljana, Slovenia
- South Africa (3):
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Mayville, KwaZulu-Natal
- Spain (4):
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Esplugues Llobregat(Barcelona)
  - Novo Nordisk Investigational Site, Leganés
  - Novo Nordisk Investigational Site, Madrid

REFERENCES:
- [Background] Thalange N, Deeb L, Klingensmith G, Franco DR, Bardtrum L, Tutkunkardas D, Danne T. The rate of hyperglycemia and ketosis with insulin degludec-based treatment compared with insulin detemir in pediatric patients with type 1 diabetes: An analysis of data from two randomized trials. Pediatr Diabetes. 2019 May;20(3):314-320. doi: 10.1111/pedi.12821. Epub 2019 Feb 10. PMID 30666772
- [Result] Battelino T, Deeb LC, Ekelund M, Kinduryte O, Klingensmith GJ, Kocova M, Kovarenko M, Shehadeh N. Efficacy and safety of a fixed combination of insulin degludec/insulin aspart in children and adolescents with type 1 diabetes: A randomized trial. Pediatr Diabetes. 2018 Nov;19(7):1263-1270. doi: 10.1111/pedi.12724. Epub 2018 Aug 16. PMID 30014589
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 63 sites in 14 countries as follows: Belgium: 3 sites; Brazil: 1 sites; Canada:
  3 sites; Czech Republic 3 sites; Croatia: 2 sites; Israel: 6 sites; Macedonia: 2 sites; Poland: 3 sites; Russia: 5 sites; Serbia: 4 sites; Slovenia: 1 sites; South Africa: 2 sites; Spain: 5 sites; and United States: 23 sites.
Groups:
- IDegAsp OD: Insulin degludec/insulin aspart (IDegAsp) once daily (OD) 2-4U was administered subcutaneously in the thigh, upper arm (deltoid area) or abdomen with the main meal and IAsp was given with the remaining meals 1-3 times daily for 16 weeks.
- IDet OD/BID: Insulin detemir (IDet) OD/BID (once daily /twice daily) 2-4U was administered subcutaneously in the thigh, upper arm (deltoid area) or abdomen with the main meal and IAsp was given with the remaining meals 2-4 times daily for 16 weeks
Period: Overall Study
Arm/Group | IDegAsp OD | IDet OD/BID
Started | 182 | 180
Exposed | 181 (One subject was withdrawn before exposure.) | 179 (One subject was withdrawn before exposure)
Completed | 174 | 168
Not Completed | 8 | 12
Not completed — Adverse Event | 1 | 0
Not completed — other | 0 | 2
Not completed — Withdrawal by Subject | 6 | 10
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis set (FAS) included all randomised subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | IDegAsp OD | IDet OD/BID | Total
Number analyzed (Participants) | 182 | 180 | 362
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.5 (4.3) | 10.8 (4.6) | 10.6 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 94 | 187
  Male | 89 | 86 | 175
HbA1c [Mean (Standard Deviation); unit: percentage (%)] | 8.1 (1.2) | 8.1 (1.2) | 8.1 (1.2)
Fasting plasma Glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] — Capillary blood samples for fasting plasma glucose (FPG) were taken either at home or at the clinic in the morning on the day of visits 2, 14 and 18 by use of a home blood sampling kit. At baseline FPG assessment: IDegAsp OD: 172 subjects, IDet: 166 subjects. In total: 338 subjects
  mmol/L | 8.6 (4.4) | 8.1 (4.2) | 8.4 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (Glycosylated Haemoglobin) (%)
Description: Percentage point change in glycosylated haemoglobin A1c (HbA1c) from baseline (week 0) to 16 Weeks. Change from baseline summary statistics at week 16 contains only those who had both baseline and week 16 assesment.
Time Frame: Week 0 to week 16
Population: The FAS included all randomised subjects. 20 subjects were withdrawn and only 4 subjects though completed the study did not have assesments.
Measure: Mean (Standard Deviation); unit: percentage (%)
Arm/Group | IDegAsp OD | IDet OD/BID
Number analyzed (Participants) | 173 | 165
percentage (%) | -0.3 (1.0) | -0.3 (0.9)

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose
Description: Change from baseline in FPG after 16 weeks of treatment. Change from baseline summary statistics at week 16 contains only those who had both baseline and week 16 assesment.
Time Frame: week 0, week 16
Population: The FAS included all randomised subjects. 338 subjects had assessment at baseline, 326 had assessment at week 16, 2 subjects were withdrawn before exposure and 22 subjects week 16 assessment was not done.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDegAsp OD | IDet OD/BID
Number analyzed (Participants) | 162 | 148
mmol/L | -0.3 (6.4) | -0.1 (4.8)

3. Secondary Outcome: Incidence of Treatment Emergent Adverse Events (TEAEs)
Description: A Treatment Emergent Adverse Event (TEAE) was defined as an event with onset date on or after the first day of exposure to randomised treatment and no later than 7 days after the last day on randomised treatment.
Time Frame: After 16 weeks of treatment
Population: The Safety analysis set (SAS) included all subjects receiving at least one dose of the trial product or its comparator
Measure: Number; unit: number of events
Arm/Group | IDegAsp OD | IDet OD/BID
Number analyzed (Participants) | 181 | 179
number of events | 501 | 460

4. Secondary Outcome: Number of Treatment Emergent Confirmed Hypoglycaemic Episodes (Plasma Glucose (PG) Below 3.1mmol/L (56mg/dL) or Severe Hypoglycaemia)
Description: Treatment emergent hypoglycaemic episodes (PG < 3.1 mmol/L (56 mg/dL) or severe hypoglycaemia).
  Confirmed hypoglycaemic episodes were defined as episodes that were either:
  1. Severe (i.e. the child is having altered mental status and cannot assist in their care, is semiconscious or unconscious or in coma with or without convulsions and may require parenteral therapy (glucagon or i.v. glucose), or
  2. An episode biochemically confirmed by PG value of <3.1 mmol/L (56 mg/dL), with or without symptoms consistent with hypoglycaemia.
Time Frame: After 16 weeks of treatment
Population: The SAS included all subjects receiving at least one dose of the trial product or its comparator
Measure: Number; unit: episodes
Arm/Group | IDegAsp OD | IDet OD/BID
Number analyzed (Participants) | 181 | 179
episodes | 2532 | 2672

5. Secondary Outcome: Number of Treatment Emergent Nocturnal Confirmed Hypoglycaemic Episodes
Description: The confirmed hypoglycaemic episodes occurring between 23:00 and 07:00 were considered for this endpoint
Time Frame: After 16 weeks of treatment
Population: The SAS included all subjects receiving at least one dose of the trial product or its comparator
Measure: Number; unit: episodes
Arm/Group | IDegAsp OD | IDet OD/BID
Number analyzed (Participants) | 181 | 179
episodes | 316 | 291

6. Secondary Outcome: Number of Hyperglycaemic Episodes (PG Above 14.0 mmol/L (250 mg/dL) Where Subject Looks/Feels Ill
Description: The episode of hyperglycaemia was noted when the glucose measurement was 14.0mmol/L or above and the subject looked /felt ill.
Time Frame: After 16 weeks of treatment
Population: The SAS included all subjects receiving at least one dose of the trial product or its comparator
Measure: Number; unit: episodes
Arm/Group | IDegAsp OD | IDet OD/BID
Number analyzed (Participants) | 181 | 179
episodes | 599 | 449

7. Secondary Outcome: Number of Hyperglycaemic Episodes (PG Above 14.0 mmol/L (250 mg/dL) Where Subject Looks/Feels Ill With Ketosis (Blood Ketones Above 1.5 mmol/L)
Description: The episode of hyperglycaemia was noted when the glucose measurement was 14.0mmol/L or above and the subject looked /felt ill. The ketone meaurement involved an additional finger prick and ketosis was considered present if blood ketones were higher than 1.5mmol/L
Time Frame: After 16 weeks of treatment
Population: The SAS included all subjects receiving at least one dose of the trial product or its comparator
Measure: Number; unit: episodes
Arm/Group | IDegAsp OD | IDet OD/BID
Number analyzed (Participants) | 181 | 179
episodes | 6 | 12

ADVERSE EVENTS:
Time Frame: Onset date on or after the first day of esxposure to randomised treatment and no later than 7 days after the last day on randomised treatment
Description: The SAS included all subjects receiving at least one dose of the trial product or its comparator
Arm/Group | IDegAsp OD | IDet OD/BID
Serious Adverse Events (participants affected / at risk) | 11/181 | 7/179
Other Adverse Events (participants affected / at risk) | 96/181 | 97/179
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegAsp OD (N=181) | IDet OD/BID (N=179)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fibula Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypoglycaemic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Developmental glaucoma (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegAsp OD (N=181) | IDet OD/BID (N=179)
Abdominal pain (Gastrointestinal disorders) | 10 (13) | 7 (13)
Abdominal pain upper (Gastrointestinal disorders) | 14 (22) | 17 (26)
Vomiting (Gastrointestinal disorders) | 22 (25) | 12 (13)
Influenza (Infections and infestations) | 9 (10) | 10 (12)
Nasopharyngitis (Infections and infestations) | 36 (43) | 32 (42)
Pharyngitis (Infections and infestations) | 3 (3) | 10 (13)
Upper respiratory tract infection (Infections and infestations) | 11 (12) | 17 (18)
Headache (Nervous system disorders) | 23 (47) | 32 (64)
Pyrexia (General disorders) | 17 (26) | 10 (15)
cough (Respiratory, thoracic and mediastinal disorders) | 13 (16) | 9 (9)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 13 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of plans by any investigator to publish and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to Novo Nordisk before submission for comments. Comments will be given within four weeks from receipt of the planned communication